CLINICAL TRIAL: NCT01638247
Title: A Prospective, Randomised, Multi-centre Phase II Study Evaluating the Adjuvant, Neoadjuvant or Palliative Treatmant With Tamoxifen +/- GnRH Analogue Versus Aromatase Inhibitor + GnRH Analogue in Male Breast Cancer Patients
Brief Title: Tamoxifen +/- GnRH Analogue vs Aromatase Inhibitor + GnRH Analogue in Male Breast Cancer Patients
Acronym: MALE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 54; 2009-015122-11 (EudraCT Number)
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Male Breast Cancer
Keywords: Male breast cancer; neoadjuvant, adjuvant or metastatic situation; anti-hormonal therapy
MeSH Terms: conditions — Breast Neoplasms, Male | interventions — Tamoxifen; Gonadotropin-Releasing Hormone; Goserelin; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tamoxifen (Active Comparator): Tamoxifen alone (daily).
  Interventions: Drug: Tamoxifen
- Tamoxifen and GnRH analogue (Experimental): Tamoxifen (daily) + GnRH analogue (at randomisation and after three months).
  Interventions: Drug: Tamoxifen and GnRH analogue
- Exemestane and GnRH analogue (Experimental): Exemestane (daily) + GnRH analogue (at randomisation and after three months).
  Interventions: Drug: Exemestane and GnRH analogue

INTERVENTIONS:
Drug: Tamoxifen — 25 mg daily.
  Arms: Tamoxifen
Drug: Tamoxifen and GnRH analogue — 25 mg Tamoxifen daily and GnRH analogue:
  * Goserelin (10.8 mg s.c. after randomisation and after three months) or
  * Leuprorelin (11.25 mg s.c. after randomisation and after three months).
  Other Names: TRENATONE, ZOLADEX
  Arms: Tamoxifen and GnRH analogue
Drug: Exemestane and GnRH analogue — 25 mg Exemestane daily and GnRH analogue:
  * Goserelin (10.8 mg s.c. after randomisation and after three months) or
  * Leuprorelin (11.25 mg s.c. after randomisation and after three months).
  Other Names: AROMASIN, TRENATONE, ZOLADEX.
  Arms: Exemestane and GnRH analogue

SUMMARY:
A prospective, randomised multi-centre phase II study evaluating the adjuvant, neoadjuvant or palliative treatment with tamoxifen +/- GnRH analogue versus aromatase inhibitor + GnRH analogue in male breast cancer patients (MALE).

DETAILED DESCRIPTION:
Breast cancer in men is a rare disease with approximately 0.5- 1% of all breast cancer cases. Each year, about 400 to 450 cases are diagnosed in Germany. Men tend to present with more advanced disease than women, probably due to the lack of awareness of male breast cancer from both, the patient and the physicians.

Therefore, at presentation they usually have lump or nipple inversion, and more than 40% of the patients have a stage III or IV disease. The great majority of patients have an invasive ductal (90%), hormone receptor positive (90%), HER2 negative (90%) tumor.

The only available information on adjuvant therapies derives from few retrospective cases and retrospective studies with a little number of cases. Therefore, treatment strategies are not based on data from prospective, randomised clinical studies, and optimal treatment is unknown. As a result, current clinical management is generally extrapolated from principles established for the treatment of female breast carcinoma. As the majority of male breast cancer patients have a hormone receptor positive tumor, they receive tamoxifen 20 mg for five years as standard endocrine adjuvant therapy. A lot of withdrawals from the treatment were documented in male breast cancer due to side-effects under tamoxifen therapy. Furthermore, the clinical outcome of tamoxifen-treated male breast cancer patients may be influenced by the activity of cytochrome P450 2D6 enzymes that catalyse the formation of anti-estrogenic metabolites endoxifen and 4-hydroxy-tamoxifen. Therefore a significant proportion of poor to moderate metaboliser is proposed to do not benefit from adjuvant tamoxifen therapy.

Although women benefit from adjuvant treatment with aromatase inhibitors (AI) regarding disease-free-survival, overall survival and treatment toxicity, only case reports of men treated with AI exist. Other data show, that under AI, there is only a suppression of estradiol of about 40-50% with an increase of testosterone of about 50%. Among men on AIs, it is possible that the hypothalamic-pituitary feedback loop results in an increase substrate for aromatisation, and thus prevents complete estrogen suppression.

However, an optimal suppression (80%) of the peripheral estradiol level would be a necessary condition for a therapeutic benefit of AI in men with breast cancer.

By adding a gonadotropin-releasing hormone analogue, the negative feedback loop would be interrupted and complete estrogen suppression may be achieved.

In conclusion, there is a great lack on information for the treatment of male patients with breast cancer.

Prospective multi-centre, randomised trials in men with breast cancer are necessary in order to prove the effect of tamoxifen + GnRH analogue versus none and versus AI + GnRH analogue as adjuvant or neoadjuvant endocrine treatment.

ELIGIBILITY:
Inclusion criteria

1. Written informed consent for all study procedures.
2. Complete baseline documentation sent to GBG Forschungs GmbH.
3. Male patients.
4. Age ≥ 18 years.
5. Karnofsky-Index ≥ 60%.
6. Histologically confirmed unilateral or bilateral carcinoma or of the breast at primary diagnosis (enrolment possible in neoadjuvant, adjuvant and metastatic situation).

7: No target lesion necessary for metastatic situation 8. Positive hormone receptor status (e.g. ER and/or PR-receptor positive). 9. Completed staging prior randomisation ( within 8 weeks after diagnose or last therapy (operation, chemotherapy or radiation), minimum: chest X-ray, ultrasound of the liver, bone scan).

In case of positive findings, further investigations are required to verify the findings as clinically indicated.

10. Prior chemotherapy is possible. In case of adjuvant treatment: adequate surgical treatment with histological complete resection including axillary lymph nodes if patients are included as adjuvant treatment. A sentinel lymph node biopsy is possible if the sentinel is not involved.

11. Normal cardiac function must be confirmed by ECG within three months prior to randomisation.

12. Laboratory requirements (≤ 14 days before therapy start): Hematology

* Hemoglobin ≥ 9 g/dL,
* Leukocytes 4 - 10 x1000/µL,
* Thrombocytes 150 - 400 x1000/µL. Hepatic function
* ASAT (SGOT) or ALAT (SGPT) ≤ 2x UNL,
* Total bilirubin ≤ 2x UNL. Renal function
* Serum creatinine ≤ 1.5x UNL,
* Creatinine clearance > 30 mL/min (if creatinine is above UNL, according to Cockroft-Gault).
* Cholesterol 200 - 240 mg/dL (5.18 - 6.22 mmol/L),
* HDL cholesterol > 40 mg/dL (> 1 mmol/L),
* LDL cholesterol ≤ 160 mg/dL (≤ 4 mmol/L).
* Prostate specific antigen (PSA) ≤ 2.5 ng/mL. 13. Two serum samples (5 mL) centrally made available. 14. Paraffin tumor tissue block and full blood sample centrally made available (except when the patient does not agree to central biomaterial collection).

  15. The patient must be accessible for treatment. Patients can simultaneously be registered in the register study of the University Hospital of Magdeburg.

Exclusion Criteria

1. Female patients.
2. Prior endocrine therapy of breast carcinoma.
3. Known or suspected hypersensitivity reaction to the compounds or incorporated substances.
4. No indication for endocrine treatment.
5. Life expectancy of less than six months.
6. International Prostate Symptom Score (IPSS) > 17.
7. Current diagnosis of a Prostate carcinoma.
8. History of prostate cancer within the last five years and regardless the time frame all patients with hormone receptor positive prostate carcinoma who have received endocrine treatment.
9. Concurrent neuronal or cardiac disease, poorly controlled arterial hypertension.
10. Previous thromboembolic event within the last five years (except from thromboembolic events correlated to implanted devices (e.g. port thrombosis)
11. Currently active hepatitis.
12. Disease significantly affecting gastrointestinal function, e.g. malabsorption syndrome, resection of the stomach or small bowel.
13. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational, not marketed drug within 30 days prior to study entry.
14. Patients who are not able to give informed consent as defined according to AMG.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Estradiol blood concentation | 3 months.
  To determine the estradiol suppression between the three treatment arms after three months.

SECONDARY OUTCOMES:
Estradiol blood concentration | 6 months.
  To determine the estradiol suppression between the three treatment arms after six months.
Compliance | 6 months.
  To compare the compliance in the three treatment arms.
Efficacy | 6 months.
  To compare the efficacy in terms of overall response (for neoadjuvant and metastatic patients) in the three treatment arms.
Efficacy perameters | 6 months.
  To compare testosterone, dihydrotestosterone (DHT), SHBG, FSH, LH, osteocalcin and CTX in the three treatments arms.
Safety and side effect parameters | 6 months.
  To determine the safety and side effect parameters (at every visit):
  * PSA and hemoglobin.
  * Lipids (total cholesterol, high density lipid cholesterol, low density lipid cholesterol).

CONTACTS AND LOCATIONS:
Overall Officials: Mattea Reinisch, MD, Principal Investigator — Kliniken Essen-Mitte
Locations (1):
- Kliniken Essen-Mitte, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Reinisch M, Seiler S, Hauzenberger T, Kamischke A, Schmatloch S, Strittmatter HJ, Zahm DM, Thode C, Furlanetto J, Strik D, Mobus V, Reimer T, Sinn BV, Stickeler E, Marme F, Janni W, Schmidt M, Rudlowski C, Untch M, Nekljudova V, Loibl S. Efficacy of Endocrine Therapy for the Treatment of Breast Cancer in Men: Results from the MALE Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 Apr 1;7(4):565-572. doi: 10.1001/jamaoncol.2020.7442. PMID 33538790
- See also: Sponsor study homepage — https://www.gbg.de/de/studien/male.php